CLINICAL TRIAL: NCT02581748
Title: A Phase I Study to Evaluate the Safety and Tolerability of Different Dosages of HLX02 (Open-label Part) and to Compare the Pharmacokinetics, Safety, Tolerability, and Immunogenicity Between HLX02 and Herceptin® (US and Germany Sourced; Double-blind, Randomized, Parallel-group Part) in Healthy Chinese Male Subjects
Brief Title: A Safety and Pharmacokinetic Study Between HLX02 and Herceptin®(U.S. and German Sourced) in Healthy Chinese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX02-HV01
Record Dates: First submitted 2015-10-09; First posted 2015-10-21 (Estimated); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Healthy
MeSH Terms: interventions — Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- safety (Experimental): Assessment of safety of HLX02 at different doses
  Interventions: Drug: HLX02
- PK comparative (Active Comparator): Randomised, double-blind, parallel group Phase I study to compare PK profiles and to assess the safety and immunogenicity between HLX02 and Herceptin®(U.S. and German)
  Interventions: Drug: HLX02; Drug: Herceptin

INTERVENTIONS:
Drug: HLX02
Drug: Herceptin
  Arms: PK comparative

SUMMARY:
Assessment of safety of HLX02 at different doses. Randomised, double-blind, parallel group Phase I study to compare PK profiles and to assess the safety and immunogenicity between HLX02 and Herceptin® (U.S. and German).

ELIGIBILITY:
Inclusion Criteria:

1. Provide the singed informed consent form (ICF)
2. Healthy Chinese male subjects (healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination including blood pressure and pulse rate measurement, 12 lead ECG, and clinical laboratory tests)
3. Aged ≥18 and ≤45 years
4. Body mass index (BMI) ≥19 and ≤28 kg/m2
5. Weight ≥50 and ≤80 kg
6. Left ventricular ejection fraction (LVEF) falls within the normal range as measured by echocardiogram (ECHO) within 14 days prior to randomisation
7. Subjects must agree that they and their female spouse/partners will use reliable contraception (2 forms of birth control, one of which must be barrier method) or be of non-childbearing potential from the time of the administration of investigational product (IP) until the completion of the study
8. Do not smoke or smoke fewer than 5 cigarettes daily within three months prior to screening; do not drink or drink less than 14 units of alcohol within six months prior to screening (1 unit of alcohol = 360 mL beer or 45 mL spirits with 40% alcohol content or 150 mL wine)

Exclusion Criteria:

1. Any history of clinically serious diseases such as hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, oncologic, or allergic diseases
2. Clinically significant abnormalities in laboratory test results
3. Previous exposure to any monoclonal antibody or current use of any biologics
4. History of allergic or anaphylactic reactions including those occurred during any clinical study or those caused by any drug or any of its excipients
5. Use of prescription or non prescription drugs and dietary supplements, within 5 half-lives of the drug or supplement, or within 2 weeks prior to taking IP (whichever is longer). Herbal supplements must be discontinued 28 days prior to the IP
6. History of a blood donation within 3 months prior to the administration of IP
7. Have participated in any other clinical study within 3 months prior to the administration of IP
8. Have positive test results for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies, or human immunodeficiency virus (HIV) antibodies
9. Have a history of drug abuse
10. Unlikely to comply with the protocol requirements, instructions, and study related restrictions; e.g., uncooperative attitude, inability to return for follow-up visits or improbability of completing the whole clinical study, etc.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2015-09-16 (Actual); Primary Completion 2016-05-11 (Actual); Study Completion 2017-01-25 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time zero to infinity (AUCinf) | 57 days

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) | 57 days
Time to Cmax (Tmax) | 57 days
Adverse event frequencies | 57 days
Area under the concentration-time curve from time zero to the last quantifiable concentration (AUClast) | 57 days

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

REFERENCES:
- [Derived] Zhu X, Ding Y, Yu Y, Wang M, Zhou W, Wang J, Zhu X, Zhang H, Wang M, Chai K, Zhang X, Luk A, Jiang W, Liu S, Zhang Q. A Phase 1 randomized study compare the pharmacokinetics, safety and immunogenicity of HLX02 to reference CN- and EU-sourced trastuzumab in healthy subjects. Cancer Chemother Pharmacol. 2021 Mar;87(3):349-359. doi: 10.1007/s00280-020-04196-9. Epub 2020 Nov 9. PMID 33169186